CLINICAL TRIAL: NCT02381301
Title: Biomarkers and Cardiac Computed Tomography: Relationship Between Cardiovascular Biomarkers and Coronary Artery Disease in Patients Undergoing Cardiac Computed Tomography
Brief Title: Biomarkers and Cardiac CT
Status: Recruiting | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: METC 14-4-117
Record Dates: First submitted 2015-03-02; First posted 2015-03-06 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease; Atherosclerosis
Keywords: Biological Markers; Multidetector Computed Tomography
MeSH Terms: conditions — Coronary Artery Disease; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Venous blood sampling prior to CCTA.: In patients undergoing routine Cardiac Computed Tomography Angiography (CCTA) and given written informed consent blood sampling will be performed. The samples will be stored for a period of 15 years at the Biobank for future analyses.
  Interventions: Biological: Venous blood sampling prior to CCTA.

INTERVENTIONS:
Biological: Venous blood sampling prior to CCTA.

SUMMARY:
Coronary artery disease (CAD) is the leading cause of morbidity and mortality in developed countries. In addition, many patients suffer from valvular and aortic disease. Although various tools are available to identify patients with cardiovascular (CV) disease at risk for major adverse cardiac events (MACE), the identification of these patients remains a clinical challenge.

One promising avenue is the use of different serum biomarkers involved in atherothrombosis which could provide an easy and cost-effective step in risk stratification.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred from the Cardiology clinic for routine CCTA.

Exclusion Criteria:

* Pregnancy
* Severe renal insufficiency
* Severe allergy to contrast medium
* Inability to obtain informed consent
* Age below 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients referred from the Cardiology clinic for routine CCTA for diagnostic purposes, will be included in this study, after given written informed consent.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-02; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Data registration of patients undergoing CCTA and given written informed consent. | 15 years.
To detect these patients for cardiovascular disease and Long term CV outcome (MACE). | 15 years.

SECONDARY OUTCOMES:
The relationship of novel blood biomarkers with CCTA findings. | 15 years.
The predictive value of these biomarkers to predict CAD in patients undergoing CCTA. | 15 years.
The prognostic value of these biomarkers (in combination) to predict MACE. | 15 years.

CONTACTS AND LOCATIONS:
Overall Officials: Harry J Crijns, MD, PhD, Study Chair — Maastricht University Medical Center; Bas Kietselaer, MD, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands